CLINICAL TRIAL: NCT04093128
Title: Beneficial Effects of Herbal Tea on Lipid Profile, Insulin Resistance, CRP, CBC, Liver, and Kidney Function Tests, and Anthropometric Indices in Jordanian Adults
Brief Title: Investigate Beneficial Effect of Herbal Tea in Jordanian Adults
Acronym: herbaltea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dr.Ruba Musharbash (Other)
Responsible Party: Sponsor-Investigator, Dr.Ruba Musharbash, Principal investigator, Ruba Musharbash Nutrition Consultancy Center
Organization: Ruba Musharbash Nutrition Consultancy Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1762019
Record Dates: First submitted 2019-07-19; First posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Diet, Healthy
Keywords: herbal tea; infusion; carob; green tea; anise; insulin resistance; inflammation; health; lipid profile; manuka honey
MeSH Terms: conditions — Insulin Resistance; Inflammation | interventions — Teas, Herbal; locust bean gum; anise oil; Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adults aged 19-57 (Experimental): adults aged 19-57 years old living in Amman Jordan, body mass index between 19-57
  Interventions: Other: herbal tea intervention

INTERVENTIONS:
Other: herbal tea intervention — herbal tea intervention for 7 weeks
  Other Names: herbal tea; carob; anise; green tea; manuka honey; wild thyme; eucalyptus leaves

SUMMARY:
investigate beneficial effect of an herbal tea prepared from carob pulp and pods (Ceratonia siliqua), anise seed (Pimpinella Anisum L), wild thyme, green tea and eucalyptus leaves with Manuka honey (natural sweetener) on lipid profile and insulin resistance, CRP (C-reactive protein), CBC (complete blood count), liver function test, kidney function tests, inflammation and anthropometric indices in adults living in Amman Jordan

DETAILED DESCRIPTION:
This study will be carried out to examine the effect of herbal tea in recruited subjects in an intervention single-group pretest-posttest study for a period of 7 weeks. Subjects will consume twice a day for a period of 7 weeks an herbal tea of (carob, anise, wild thyme, and eucalyptus leaves) before eating. The total sample (n=30) adults aged (19-57 years) , body mass index BMI range (19-35 kg/m2)

ELIGIBILITY:
Inclusion Criteria:

* adults aged 19-57 years
* male to female ratio (1:1 ratio)
* BMI 19-35 kg/m2
* Currently living in Amman
* without significant apparent diseases
* Able to drink the tested herbal tea twice a day

Exclusion Criteria:

* Have chronic diseases such as diabetes, hypertension, cardiovascular or endocrine diseases or disabilities
* Using medical drugs and/or supplements
* Below 19 or above 57 years.
* participation in clinical trials within the last 2 months
* use of lipid-lowering drugs, or diabetic medication.
* Lactating and pregnant women will be also excluded.

Ages: 19 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
Questionnaire | 1-2 weeks
  basic demographic information
Homocysteine serum level | 7 weeks pre and post intervention
  venous blood sample for 30 candidates measured by umol/L normal range < 12 umol/L
Fasting blood sugar | 7 weeks pre and post intervention
  venous blood sample for 30 candidates measured by mg/dL normal range 70-99 mg/dL
Glycosylated Haemoglobin (HBA1C) blood | 7 weeks pre and post intervention
  venous blood sample for 30 candidates measured by percentage normal range 4.8-5.8%
Cholesterol serum | 7 weeks pre and post intervention
  venous blood sample for 30 candidates measured by mg/dL normal range <200 mg/dL
Triglyceride serum | 7 weeks pre and post intervention
  venous blood sample for 30 candidates measured by mg/dL normal range <150 mg/dL
HDL cholesterol(High density lipoprotein) serum | 7 weeks pre and post intervention
  venous blood sample for 30 candidates measured by mg/dL normal range >60mg/dL
Cholesterol/HDL Ratio | 7 weeks pre and post intervention
  venous blood sample for 30 candidates normal range <4.0
LDL Cholesterol (low density lipoprotein) serum | 7 weeks pre and post intervention
  venous blood sample for 30 candidates measured by mg/dL normal range <100mg/dL
Protein serum | 7 weeks pre and post intervention
  venous blood sample for 30 candidates measured by g/dL normal range 6.0-8.0g/dL
C-Reactive Protein high sensitivity serum | 7 weeks pre and post intervention
  venous blood sample for 30 candidates measured by mg/dL , low risk of CVD <1.0 mg/dL
Insulin serum | 7 weeks pre and post intervention
  venous blood sample for 30 candidates measured by uU/ml normal range 2.6-24.9
Cortisol Total (AM) serum | 7 weeks pre and post intervention
  venous blood sample for 30 candidates measured by ug/dL normal range 6.02-18.4
Tumor Necrosis Factor | 7 weeks pre and post intervention
  venous blood sample for 30 candidates measured by pg/mL normal range upto 8.1
8-OH-2 Desoxyyguanosine urine | 7 weeks pre and post intervention
  Urine sample measured by micromol/mol normal range 0.1-2.4
interleukin 1 Beta | 7 weeks pre and post intervention
  venous blood sample for 30 candidates measured by pg/ml normal range upto 5 pg/ml
weight | 7 weeks pre and post intervention
  measured on inbody 770 measured by kg
Height | pre intervention
  measured by cm

SECONDARY OUTCOMES:
gastrointestinal symptoms questionnaire | 7 weeks pre and post intervention
  measure severity of GI symptoms including bloating , flatulence, gastrointestinal pain and loss of appetite, measure the occurrence of these symptoms and reduction in mean severity symptoms after herbal intervention
Creatinine serum | 7 weeks pre and post intervention
  venous blood sample for 30 candidates measured by mg/dL normal range male 0.7-1.2mg/dL females 0.5-0.9mg/dL
Alanine Aminotransferase (ALT/GPT) serum | 7 weeks pre and post intervention
  Venous blood sample for 30 candidates measured by U/L normal range Upto 41 U/L
Aspartate Aminotransferase (AST/GOT) serum | 7 weeks pre and post intervention
  Venous blood sample for 30 candidates measured by U/L normal range Upto 40 U/L
Gamma-Glutamyl Transferase (GGT) serum | 7 weeks pre and post intervention
  Venous blood sample for 30 candidates measured by U/L normal range 8-61 U/L
Alkaline phosphatase serum | 7 weeks pre and post intervention
  Venous blood sample for 30 candidates measured by U/L normal range 40-129
Creatine phospho Kinase (CPK) | 7 weeks pre and post intervention
  Venous blood sample for 30 candidates measured by U/L normal range males 20-200 U/L females 20-180 U/L
Microalbuminuria spot urine | 7 weeks pre and post intervention
  Urine sample measured by mg/L normal range <20.0 mg/L
Creatinine spot urine | 7 weeks pre and post intervention
  Urine sample measured by mg/dL normal range males 39-259 mgd/L females 28-217mg/dL
Microalbuminuria-Creatinine spot urine | 7 weeks pre and post intervention
  Urine sample measured by by mg/g creat. normal range < 30.0 mg/g creat.
Haemoglobin | 7 weeks pre and post intervention
  Venous blood sample for 30 candidates measured by gm/L males 140-180 gm/L females 120-160 gm/L
haematocrit | 7 weeks pre and post intervention
  Venous blood sample for 30 candidates measured by L/L males 0.42-0.54L/L females 0.37-0.47 L/L
Erythrocytes | 7 weeks pre and post intervention
  Venous blood sample for 30 candidates measured by x10^12/L males 4.7-6.1 x10^12/L females 4.2-5.4 x10^12/L
MCV | 7 weeks pre and post intervention
  Venous blood sample for 30 candidates measured by FL normal range 80-96 FL
MCH | 7 weeks pre and post intervention
  Venous blood sample for 30 candidates measured by pg normal range 27-31 pg
MCHC | 7 weeks pre and post intervention
  Venous blood sample for 30 candidates measured by gm/L normal range 320-360gm/L
RDW- cv | 7 weeks pre and post intervention
  Venous blood sample for 30 candidates measured by percentage normal range 11.5-14.5%
Leukocytes | 7 weeks pre and post intervention
  Venous blood sample for 30 candidates measured by x10^9/L normal range 4.500-10.000
platelets | 7 weeks pre and post intervention
  Venous blood sample for 30 candidates measured by x10^9/L normal range 150-400
Skeletal muscle mass | 7 weeks pre and post intervention
  measured on inbody 770 measured by kg
Body fat mass | 7 weeks pre and post intervention
  measured on inbody 770 measured by kg
Percent body fat mass | 7 weeks pre and post intervention
  measured on inbody 770 measured by percentage
free fat muscle | 7 weeks pre and post intervention
  measured on inbody 770 measured by kg
Visceral fat are | 7 weeks pre and post intervention
  measured on inbody 770 measured by cm2
total body water | 7 weeks pre and post intervention
  measured on inbody 770 measured by L
Body mass index | 7 weeks pre and post intervention
  measured on inbody 770 measured by kg/m2
Basal metabolic rate | 7 weeks pre and post intervention
  measured on inbody 770 measured by kcal
waist circumference | 7 weeks pre and post intervention
  measured by cm measures using measuring tape
Hip circumference | 7 weeks pre and post intervention
  measured by cm measures using measuring tape
Waist/hip ratio | 7 weeks pre and post intervention
  measured using equation waist/hip
Waist/height ratio | 7 weeks pre and post intervention
  measured using equation waist/height

CONTACTS AND LOCATIONS:
Locations (1):
- Ruba Musharbash, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No